CLINICAL TRIAL: NCT06121869
Title: A Pilot Study to Examine Changes in Resistance Training Adaptations After Leucine and Dileucine Ingestion
Brief Title: Dileucine and Resistance Training Adaptations
Acronym: DTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Collaborators: Ingenious Ingredients, L.P. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-41-64
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Hypertrophy; Strength Training Adaptations; Weight-Bearing Strengthening Program
Keywords: Peptides; Dipeptide; Adaptations; Exercise; Dietary Supplements
MeSH Terms: conditions — Hypertrophy; Motor Activity | interventions — Leucine

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator
Masking Description: All supplements will be provided in blinded, labeled containers prior to them arriving to the site. Each supplement will be of similar volume, texture, and labeled in indistinguishable bottles to ensure blinding of both participant and invesitigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will supplement daily for 10 weeks with 2 grams rice flower placebo in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Interventions: Dietary Supplement: Placebo
- Leucine (Active Comparator): Participants will supplement daily for 10 weeks with 2 grams rice leucine in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Interventions: Dietary Supplement: Leucine
- Dileucine (Experimental): Participants will supplement daily for 10 weeks with 2 grams dileucine (RAMPS, Ingenious Ingredients, TX, USA) in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Interventions: Dietary Supplement: Dileucine

INTERVENTIONS:
Dietary Supplement: Placebo — Participants will supplement daily for 10 weeks with 2 grams rice flower placebo in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Arms: Placebo
Dietary Supplement: Leucine — Participants will supplement daily for 10 weeks with 2 grams leucine in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Arms: Leucine
Dietary Supplement: Dileucine — Participants will supplement daily for 10 weeks with 2 grams dileucine (RAMPS, Ingenious Ingredients, TX, USA) in capsule form. On training days, participants will consume their assigned supplement within 60 minutes of completing their workout. On non-training days, participants will consume their assigned supplement with their first meal of the day. All doses will be consumed with 8-12 ounces of water.
  Arms: Dileucine

SUMMARY:
This study seeks to compare the observed changes in resistance training adaptations after supplementation of isomolar amounts of leucine or dileucine in healthy resistance-trained men. This will provide a better understanding of supplementation with leucine versus dileucine over a 10-week period in regards to increasing muscular performance.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind approach with individuals being provided daily 2-gram doses of leucine, 2-gram doses of dileucine, or a placebo. Daily blinded supplementation will occur each day for a 10-week period of time while completing a heavy resistance training program. Participants follow the resistance training program for a total of 10 weeks. To compare the efficacy of leucine in form of amino acid or dipeptide supplementation on resistance training adaptations, changes in fat-free, lean, and fat mass will be determined using a 4-compartment body composition model. Skeletal muscle cross-sectional area will be assessed using ultrasound. Maximal strength, muscular endurance, and power will also be assessed. Participants will be required to provide weekly compliance and complete one supervised workout per week. After 2, 6, and 10 weeks of following the supplementation and resistance training regimens, participants will return to the laboratory to complete testing bouts consisting of identical assessments of body composition, muscular strength, muscular endurance, lower-body power, and anaerobic capacity. Adverse events related to each supplementation group will be recorded and assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between the ages of 18-39 years of age
* Currently participating in resistance training exercise

Exclusion Criteria:

* Female
* Participants who are determined to not be weight stable defined as week 0 and week 2 body mass levels deviating by 3% or more.
* Any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, immune, autoimmune, psychiatric, hematological, neurological or endocrinological disorder or disease.
* Body mass index > 25 kg/m2. Individuals with a body mass index greater than 25 kg/m2, but a body fat percentage less than 25% fat will be accepted into the study
* Individuals who present with any previous injury or illness that would prevent them from appropriately completing all exercise lifts.
* Participants who are not able to fit onto the DEXA table will not be able to participate in the research due to size restrictions of the equipment. This typically includes individuals exceeding 400 pounds or those greater than 6'4".
* Those individuals with less than 12 months of structured resistance training experience will be excluded from the study.
* Individuals whose maximal relative upper body strength is below 1.0 will be excluded.
* Individuals whose maximal relative lower body strength is below 1.5 will be excluded.
* All participants who DO NOT abstain from taking any additional forms of nutritional supplementation deemed to be ergogenic or that will impact resistance training adaptations (pre-workouts, creatine, beta-alanine, etc.) for four weeks prior to beginning this study and for the entire duration of the study.
* Individuals who are currently using or have used within the past 12 months anabolic-androgenic steroids.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Fat-Free Mass | 10 weeks
  Fat-free mass will be determined via Dual-Energy X-Ray Absorptiometry
Leg Press 1RM | 10 weeks
  Leg Press 1RM will be measured using the leg press (lower-body) exercise.
Bench Press 1RM | 10 weeks
  Bench Press 1RM will be measured using the bench press (upper-body) exercise.
Maximal Isometric Mid-Thigh Pull Force Production | 10 weeks
  Maximal Isometric Mid-Thigh Pull Force Production will be measured using an isometric mid-thigh pull test

SECONDARY OUTCOMES:
Fat Mass | 10 weeks
  Fat mass will be determined via Dual-Energy X-Ray Absorptiometry
Lean mass | 10 weeks
  Lean mass will be determined via Dual-Energy X-Ray Absorptiometry
% Body Fat | 10 weeks
  % Body Fat will be determined via Dual-Energy X-Ray Absorptiometry
Total body water | 10 weeks
  Total Body Water will be determined via bioelectrical impedance analysis
Extracellular Body Water | 10 weeks
  Extracellular Body Water will be determined via bioelectrical impedance analysis
Intracellular Body Water | 10 weeks
  Intracellular Body Water will be determined via bioelectrical impedance analysis
Skeletal muscle cross-sectional area | 10 weeks
  Skeletal muscle cross-sectional area will be measured using ultrasound measurements of the participants thigh muscles.
Bench Press Repetitions to Fatigue | 10 weeks
  Bench Press repetitions to fatigue will be measured using the bench press (upper-body) exercises on four separate occasions (visits 2, 3, 4, and 5). To complete this assessment, study participants will use a load that corresponds to 80% of their Visit 2 1RM for bench press exercise and will be instructed to complete as many repetitions as they can until failure for one set of each exercise. Failure will be defined as resting for more than two seconds throughout any point on the exercise set or technique failure.
Leg Press Repetitions to Fatigue | 10 weeks
  Leg Press repetitions to fatigue will be measured using the leg press (lower-body) exercises on four separate occasions (visits 2, 3, 4, and 5). To complete this assessment, study participants will use a load that corresponds to 80% of their Visit 2 1RM for leg press exercise and will be instructed to complete as many repetitions as they can until failure for one set of each exercise. Failure will be defined as resting for more than two seconds throughout any point on the exercise set or technique failure.
Peak Anaerobic Power | 10 weeks
  Peak Anaerobic Power will be measured using a Wingate Anaerobic Test lasting 30-seconds at a load set to 7.5% of week 0 body mass
Mean Anaerobic Power | 10 weeks
  Mean Anaerobic Power will be measured using a Wingate Anaerobic Test lasting 30-seconds at a load set to 7.5% of week 0 body mass
Rate of Fatigue | 10 weeks
  Rate of Fatigue will be measured using a Wingate Anaerobic Test lasting 30-seconds at a load set to 7.5% of week 0 body mass
Maximal Concentric Rate of Force Development | 10 weeks
  Maximal concentric rate of force development will be measured using a countermovement jump performed on a force plate

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers

REFERENCES:
- [Derived] Hagele AM, Krieger JM, Gaige CJ, Holley KF, Gross KN, Iannotti JM, Allen LE, Sutton PJ, Orr LS, Mumford PW, Purpura M, Jager R, Kerksick CM. Dileucine ingestion, but not leucine, increases lower body strength and performance following resistance training: A double-blind, randomized, placebo-controlled trial. PLoS One. 2024 Dec 31;19(12):e0312997. doi: 10.1371/journal.pone.0312997. eCollection 2024. PMID 39739679